CLINICAL TRIAL: NCT04046120
Title: Comparison of the Effectiveness of Two Medical Compression Bandage Application Techniques by Measuring Interface Pressures Depending on Whether or Not the Heel is Included in Patients With Open Venous Ulcers: Non-inferiority, Controlled, Randomized Trial
Brief Title: Comparison of the Effectiveness of Two Medical Compression Bandage Application Techniques by Measuring Interface Pressures Depending on Whether or Not the Heel is Included in Patients With Open Venous Ulcers
Acronym: COMPARACHILLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC19_0072
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Venous Ulcer
Keywords: varicose ulcer; compression bandages; patient compliance; heel; methods
MeSH Terms: conditions — Varicose Ulcer; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heel included (No Intervention): The bandage is made by including the heel as recommended in routine.
- Heel not included (Experimental): he bandage is made by leaving the heel uncovered.
  Interventions: Other: Heel-free bandage

INTERVENTIONS:
Other: Heel-free bandage — The bandage is made by leaving the heel uncovered.
  Arms: Heel not included

SUMMARY:
The importance of wearing medical compression to heal the venous ulcer has already been shown. However, no studies have been carried out on variations in medical compression tape and their impact on interface pressures which explains the lack of consensus on how to lay, including or not to include the heel. Studies on adherence to patients with medical compression have been carried out showing that one of the determining factors is comfort. The investigators therefore wish to conduct a randomized open prospective quantitative study comparing these two modes: including or not the heel .

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patient with at least one venous ulcer progressing for at least 4 weeks
* Patient coming for a specialized outpatient consultation called "vascular wound" at Nantes University Hospital
* Informed consent to participate in the study
* Social security insurance affiliation

Exclusion Criteria:

* Patients under guardianship
* Patient with major cognitive disorders incompatible with follow-up of protocol
* Pregnancy
* Patient with an open leg ulcer with a Systolic Pressure Index < 0.8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Interface pressure V3 | 48 hours after the bandage is applied (between week 4 and week 6)
  Compare the interface pressure measurements generated by a medical compression bandage between two groups of patients with open venous ulcer(s) :
  * experimental group: uncovered heel
  * control group: heel covered by the bandage.

SECONDARY OUTCOMES:
Ankle circumference | Day 0 and the last day (between week 4 and week 6)
  Compare the evolution or appearance of an edema in the ankle. The circumference of the ankle is measured with a tape measure using a technique called the figure of 8.
Interface pressure V2 | 48 hours before the last visit of the protocol. (Between 4 and 6 weeks)
  Compare, between the two groups, the interface pressures measured during the installation of bandage at home by the home nurse (V2 follow-up visit), compared to the recommended pressures (30-40 mmHg)
Interface pressure V2 and V3 | 48 hours before the last visit of the protocol and at the last visit of the protocol (Between 4 and 6 weeks)
  Compare, between the two groups, the evolution of interface pressures after 48 hours of bandage wear.
Patient satisfaction: questionnaire | At the last visit of the protocol (Between 4 and 6 weeks)
  Between the two groups, compare patient satisfaction with a heterogeneous questionnaire.
  There is no scale or score. It is asked which type of bandage the patient prefers: with or without heel included?
Number of bandage repairs | Day 0
  Evaluate the number of bandage repairs required to reach the recommended therapeutic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Anne POTTIER, Principal Investigator — Nantes University Hospital
Locations (1):
- Chu de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No